CLINICAL TRIAL: NCT04317131
Title: The Interdependence of Body Posture and the Stomatognathic System of School-age Children in Structural and Functional Terms
Brief Title: Body Posture and the Stomatognathic System of School-age Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Justyna Leszczak, PhD, University of Rzeszow
Other Study IDs: BodyPostureTMD
Record Dates: First submitted 2019-12-09; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Postural; Defect; Stomatognathic System Abnormalities; Malocclusion
Keywords: body posture; stomatognathic system; malocclusion; children
MeSH Terms: conditions — Stomatognathic System Abnormalities; Malocclusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Research Diagnostic Criteria of Functional Disorders of the Masticatory System BKD / ZCURNŻ - Polish version — Interview and clinical examination of stomatognathic system based on standardized tool BDK/ZCURNŻ.
Device: Clinical examination of the stomatognathic system (structural and functional) — Examination with the use of JMA+Analyser (Jaw Motion Analyser) to analyse movement and function of the temporomandibular joints, mandibular position, condyle position (EPA), and access the muscle action potentials through bipolar skin surface electrodes EMG, assessment of occlusion by visual method according to Angle Classification.
Device: 3D examination of the body posture — Comprehensive, three- dimensional examination of the body posture (static and dynamic) in the area of the spine, lower limbs and feet, performed by photogrammetric method (4th Generation MORA) and non- invasive image acquisition technology with the aid of infrared (Kineod) and The CQElektronik system.
Device: Functional assessment of the spine and lower limbs — Functional assessment of the spine and lower limbs mobility trough a wireless motion sensor Moover.
Device: Complementary tests — Anthropometric measurements (height, weight, waist and hip circumference, skin folds), foot pressure on the ground and body balance accessed by pedobarograph FreeMed, body mass components measured by the Tanita MC 980 MA (BIA method), evaluation of 7-days of physical activity by accelerometer ActiGraph GT3X-BT, blood pressure measurement by Medel Connect Cardio MB 10 monitor.

SUMMARY:
The aim of the study is to demonstrate a correlation between body posture and the structure and function of the stomatognathic system in school-age children.

DETAILED DESCRIPTION:
Both disorders of the stomatognathic system and body posture defects concern an increasingly younger population in Poland and in the world. The scale of both problems is constantly increasing. Structural and functional disorders in the area of the stomatognathic system have begun to be known as a disease of modern civilization. Bite defects immediately after tooth decay are the second most common dental problem for children around the world. The scale of the problem according to some sources makes up 75% of this population. Similarly, in the case of body posture defects in the spine, lower limbs and feet, it is estimated that they are present in up to 60-70% of Polish children. The critical period for the development of defects in both posture and the orofacial area falls at the same age, i.e. early school and puberty. Despite of the extensive literature describing both issues, there is still no clear and objective scientific evidence that would confirm the correlation of the two phenomena.

The presented project is an original cross-sectional study. A 400 school-age children between 6 and 15 years of age will participate in the study. Research will be conducted in randomly selected orthodontic clinics and primary schools.

The subjects will be divided into subgroups: a) children with correct body posture and without stomatognathic system dysfunction; b) children with a diagnosis of body posture defect; c) children with a diagnosis of malocclusion; d) children with a stomatognathic system dysfunction. After obtaining the mandatory written consent of the parent and child, the child's medical qualification to participate in the study will include the exclusion of: congenital structural defects of the spine, chronic diseases of the nervous system, genetic diseases, neuromuscular dystrophy, endocrine disorder, an ongoing contagious disease, present locomotor fracture, current muscular injury. The inclusion criterion will include: age of study participant from 6 to 15 years of age, in case of an existing defect in body posture/or malocclusion/or dysfunction of the stomatoghnatic system, lack of specific causes.

Methods

* interview based on standardized questionnaires, i.e. Research Diagnostic Criteria of Functional Disorders of the Masticatory System BKD / ZCURNŻ
* Polish version, TMD Questionnaire, Neck Disability Index, International Physical Activity Questionnaire (IPAQ) (short version), Questionnaire on Food Related Behavior (KZZJ)
* clinical examination of the stomatognathic system (structural and functional), using JMA+ Analyser (Jaw Motion Analyzer) to analyse movement and function of the temporomandibular joints, mandibular position, condyle position (EPA), and access the muscle action potentials through bipolar skin surface electrodes EMG, assessment of occlusion by visual method according to Angle classification.
* comprehensive 3D examination of the body posture (static and dynamic) in the area of the spine, lower limbs and feet, performed by photogrammetric method (4th Generation MORA) and non- invasive image acquisition technology with the aid of infrared (Kineod) and The CQ Elektronik system.
* functional assessment of the spine and lower limbs mobility trough a wireless motion sensor Moover.
* complementary tests, i.e. anthropometric measurements (height, weight, waist and hip circumference, skin folds), foot pressure on the ground and body balance accessed by pedobarograph FreeMed, body mass components measured by the Tanita MC 980 MA (BIA method), evaluation of 7-days of physical activity by accelerometer ActiGraph GT3X-BT, blood pressure measurement by Medel Connect Cardio MB 10 monitor.

ELIGIBILITY:
Inclusion Criteria:

* age of study participant from 6 to 15 years of age
* in case of an existing defect in body posture, lack of specific causes
* in case of an existing malocclusion, lack of specific causes
* in case of dysfunction of the stomatognathic system, lack of specific causes

Exclusion Criteria:

* congenital structural defects of the spine,
* chronic diseases of the nervous system,
* genetic diseases,
* neuromuscular dystrophy,
* endocrine disorder
* an ongoing contagious disease
* present locomotor fracture
* current muscular injury

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: A 400 school-age children between 6 and 15 years of age will participate in the study.
  Research will be conducted in randomly selected orthodontic clinics and primary schools.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-01-05 (Estimated)

PRIMARY OUTCOMES:
Clinical examination of the stomatognathic system (structural) | at baseline, immediately after medical qualification to the study
  Assessment of occlusion by visual method according to Angle classification. Research Diagnostic Criteria of Functional Disorders of the Masticatory System.
Comprehensive body posture assessment | at baseline, immediately after medical qualification to the study
  Static and dynamic body posture test using 4th Generation MORA which enables a detailed and spatial analysis of body posture by photogrammetric.
Clinical examination of the stomatognathic system (functional) | at baseline, immediately after medical qualification to the study
  JMA+ Analyser (Jaw Motion Analyzer) system will allow to analyse movement and function of the temporomandibular joints, mandibular position, condyle position (EPA), and access the muscle action potentials through bipolar skin surface electrodes EMG.
Comprehensive body posture assessment | at baseline, immediately after medical qualification to the study
  Next device used to to the body posture assessment will be KINEOD with pedobarograph which is a modern device for 3D analysis of body posture, in particular the back, but also lower limbs. The KINEOD system uses image acquisition technology with the aid of infrared. Therefore, it is a perfect complement to examining body posture using the so-called photogrammetric method, so-called moire projection method.

SECONDARY OUTCOMES:
Functional assessment of the spine and lower limbs | at baseline, immediately after medical qualification to the study
  The assessment with the use of 3D device which is intertial sensor of movement. Its application in the scientific sphere allows the goniometric evaluation (range of movement) of the articulations. In the study it allows to assess the functional head and neck mobility and additionally in lumbar spine and lower limbs joints
Anthropometric measurements | at baseline, immediately after medical qualification to the study
  Seca 213 stadiometer - equipment necessary to examine the basic anthropometric measurements of height and weight. Waist and hip circumference will be measured by centimetre tape.
Body mass composition analysis | at baseline, immediately after medical qualification to the study
  Tanita MC 780 MA- segment body mass composition analyser using the bioimpedance method (BIA). The equipment has 8 electrodes for a detailed analysis with segment reading - the division of fat and muscle mass in the left and right arm, left and right leg and body, as well as between the leg muscularity index, segment index for fat tissue and muscle mass.
Foot pressure | at baseline, immediately after medical qualification to the study
  FreeMed Posture MAXI60 Pedobarograph will allow to access pressure fields acting between the plantar surface of the foot and a supporting surface. The device shows exactly degree of patient's foot presses on the ground. Additionally, it will allow testing the patient's equivalent responses.
Body balance | at baseline, immediately after medical qualification to the study
  FreeMed Posture MAXI60 Pedobarograph will allow to access pressure fields acting between the plantar surface of the foot and a supporting surface. The device shows exactly degree of patient's foot presses on the ground. Additionally, it will allow testing the patient's equivalent responses.
7-day physical activity | at baseline, immediately after medical qualification to the study
  ActiGraph GT3X-BT accelerometers are currently the most accurate and objective motion sensors for assessing physical activity. The devices detect the acceleration of body movement in three planes, giving the possibility of reliable measurement of the intensity and duration of physical activity, as well as the number of steps performed and the time spent passively. Motion parameters are read thanks to a piezoelectric sensor. The subject will wear an accelerometer on his waist for an uninterrupted period of 7 days, excluding bathing time and swimming lessons.
Blood pressure | at baseline, immediately after medical qualification to the study
  Medel Connect Cardio MB 10 blood pressure monitor for measuring systolic and diastolic blood pressure, heartbeat values, and ECG. Each subject will have their blood pressure tested three times.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rzeszów, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: No